CLINICAL TRIAL: NCT05005234
Title: An Open-label, Multi-center Phase I/II Clinical Study Evaluating the Safety/Tolerability, Pharmacokinetics, and Effectiveness of GFH925 in Patients With Advanced Solid Tumors With KRAS G12C Mutations
Brief Title: A Study of GFH925 in Patients With Advanced Solid Tumors With KRAS G12C Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH925X1101
Record Dates: First submitted 2021-08-08; First posted 2021-08-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: KRAS G12C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFH925 (Experimental): Phase Ia Dose Escalation Subjects with advanced NSCLC and gastrointestinal tumors will be enrolled in dose escalation cohorts based on Bayesian optimal interval (BOIN) design.
  Phase Ia Dose Expansion Upon completing the dose exploration part of the study and depending on data obtained, dose expansion may proceed with responsive groups consisting of subjects with KRAS G12C mutant advanced NSCLC. Dose expansion may be done concurrently.
  Phase Ib Subjects with KRAS G12C mutant advanced colorectal cancer or other tumors will be enrolled and treated at the monotherapy RP2D to evaluate the efficacy.
  Phase 2 Subjects with KRAS G12C mutant advanced NSCLC will be enrolled and treated at the monotherapy RP2D to evaluate the safety and efficacy.
  Interventions: Drug: GFH925

INTERVENTIONS:
Drug: GFH925 — Administered as an oral tablet formulation

SUMMARY:
Phase Ia:

To evaluate the safety/tolerability of GFH925 in subjects with KRAS G12C-mutated advanced solid tumors; To estimate the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of GFH925.

Phase Ib:

To evaluate the efficacy of GFH925 in subjects with KRAS G12C mutant advanced colorectal cancer or other tumors.

Phase II:

To evaluate the efficacy of GFH925 in subjects with KRAS G12C mutant advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study and sign the informed consent form.
2. Aged 18 years or older at the time of signing the informed consent form.
3. Subjects must have one measurable lesion (per RECIST 1.1).
4. Subjects with toxic reaction caused by prior anticancer therapy need to have recovered to baseline level (except residual alopecia) or ≤ Grade 1 (neurotoxicity ≤ Grade 2 acceptable).
5. Eastern Cooperative Oncology Group (ECOG) performance status score (PS) 0 ~ 1.
6. Expected survival ≥ 12 weeks.
7. Female subjects or male subjects of childbearing potential must take effective contraceptive measures from the time of signing the informed consent form to 30 days after the last dose of GFH925, or to 60 days after the last dose of cetuximab. Female subjects of childbearing potential should have a negative blood pregnancy test within 7 days (inclusive) prior to initiation of study treatment.
8. The investigators deem the subject able to communicate well, attend regular follow-up visits, and complete the study according to the protocol.

Exclusion Criteria:

1. Significant cardiovascular system disease.
2. Subjects with unstable brain metastases diagnosed by investigators.
3. Significant gastrointestinal diseases, such as intractable hiccup, nausea, vomiting, severe gastrointestinal ulcers, cirrhosis, active gastrointestinal bleeding, or other diseases that affect swallowing tablets or significantly affect oral drug absorption; subjects with severe portal hypertension caused by the presence of Budd-Chiari syndrome or portal emboli in subjects with liver cancer also need to be excluded.
4. Presence of serious acute or chronic infections.
5. Pregnant or lactating women.
6. Known allergy to the study drug or any component of its formulation.
7. Other conditions that the investigators consider inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Phase Ia: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs); changes in laboratory tests, vital signs, physical examinations, electrocardiograms (ECGs) | Baseline to 24 Months
  Safety measures
Phase Ia: Incidence of dose-limiting toxicity (DLT) events | At the end of Cycle 1（each cycle is 21 days）
  Safety measures
Phase Ib: ORR per RECIST 1.1 | Continuous evaluation during treatment
  Efficacy measures
Phase II: ORR assessed by Independent Radiographic Review Committee (IRRC) according to RECIST 1.1 | Continuous evaluation during treatment
  Efficacy measures

SECONDARY OUTCOMES:
Phase Ia: PK parameters of GFH925 include but are not limited to: Cmax, Tmax, AUC, t1/2, CL/F and Vd/F | To complete 3 treatments cycles（each cycle is 21 days）
  Efficacy measures and safety measures
Phase Ia: Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, disease control rate (DCR), duration of response (DoR), time to response (TTR), progression-free survival (PFS),Overall survival (OS) | Continuous evaluation during treatment
  Efficacy measures
Phase Ib and Phase II: DCR, DoR, TTR, PFS per RECIST 1.1, progression-free survival rate at 6 and 12 months, overall survival rate at 12 months | Continuous evaluation during treatment
  Efficacy measures
Phase Ib and Phase II: Incidence and severity of AEs, SAEs, AEs leading to treatment interruption, and AEs leading to treatment discontinuation of GFH925 monotherapy | Baseline to 24 Months
  Safety measures
Phase Ib and Phase II: Plasma concentration (including Ctrough) after multiple dose administration in subjects | To complete 3 treatments cycles（each cycle is 21 days）
  Efficacy measures and safety measures

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No